CLINICAL TRIAL: NCT01543984
Title: Efficacy of "Tailored Physical Activity" on the Number of Sick Days: a Randomized Controlled Trial in Health Care Workers That Have Experienced Pain Related to the Spine or Upper Body
Brief Title: Efficacy of "Tailored Physical Activity" in Health Care Workers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Municipality of Sønderborg (Unknown)
Responsible Party: Principal Investigator, Lotte Nygaard Andersen, Ph.d. fellow, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 95-154-32028T
Record Dates: First submitted 2012-02-27; First posted 2012-03-05 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2014-04

CONDITIONS: Pain
Keywords: health care workers; tailored physical activity; prevention; spine; upper body; pain related to Spine or Upper body
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored Physical Activity (Experimental): Health guidance (1,5h) and "Tailored Physical Activity" (3*50 min/week in 10 weeks)
  Interventions: Other: Tailored Physical Activity
- Reference group (Other): Health Counselling (1,5h)
  Interventions: Behavioral: Health Counselling

INTERVENTIONS:
Other: Tailored Physical Activity — Tailored Physical Activity (3*50 min/week in 10 weeks)
  Arms: Tailored Physical Activity
Behavioral: Health Counselling — Health guidance (1,5h)
  Arms: Reference group

SUMMARY:
The purpose of this study is to test the effect of "Tailored Physical Activity" on the number of sick-days.

The hypothesis is that "Tailored Physical Activity" is superior in efficacy on sick-days.

DETAILED DESCRIPTION:
Health care workers have high prevalence of musculoskeletal pain. Pain in the back and neck and other musculoskeletal disorders are the leading cause for long-term sick leave.

This study test the effect of "Tailored Physical Activity" on self-reported days on sick leave and parameters regarding pain, function and quality of life respectively on the body function and participation level of health care workers which have experienced musculoskeletal pain related to the back or upper body.

A minimum of 44 health care workers in DK-Sønderborg Municipality will be randomized for "Tailored Physical Activity" or a reference group.

Primary endpoint is 3 months and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

Health care workers in municipality of Sønderborg that have experienced musculoskeletal pain related to the spine or upper body.

Exclusion Criteria:

Medically safety.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Self-reported number of sick-days | 3 months
  "How many days have you in total been on sick leave because of musculoskeletal troubles (such as ache, pain, discomfort)during the last three months" ((0 days, 1-7 days, 8-30 days, 30 days).

SECONDARY OUTCOMES:
Aerobic capacity | 3 months
Hand-grip strength | 3 months
Body weight, waist circumference, hip circumference | 3 months
Questionnaire | 3 months
Self-reported number of sick-days | 12 months follow-up
  "How many days have you in total been on sick leave because of musculoskeletal troubles (such as ache, pain, discomfort)during the last three months" ((0 days, 1-7 days, 8-30 days, 30 days).
Aerobic capacity | 12 months follow-up
Hand-grip strength | 12- months follow-up
Body weight, waist circumference, hip circumference | 12 months follow-up
Questionnaire | 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Nygaard Andersen, cand.scient, Principal Investigator — University of Southern Denmark
Locations (1):
- Health Care Centre, Sønderborg, Denmark

REFERENCES:
- [Derived] Andersen LN, Juul-Kristensen B, Roessler KK, Herborg LG, Sorensen TL, Sogaard K. Efficacy of 'Tailored Physical Activity' on reducing sickness absence among health care workers: A 3-months randomised controlled trial. Man Ther. 2015 Oct;20(5):666-71. doi: 10.1016/j.math.2015.04.017. Epub 2015 May 2. PMID 25983237
- [Derived] Andersen LN, Juul-Kristensen B, Roessler KK, Herborg LG, Sorensen TL, Sogaard K. Efficacy of 'Tailored Physical Activity' in reducing sickness absence among health care workers: design of a randomised controlled trial. BMC Public Health. 2013 Oct 2;13:917. doi: 10.1186/1471-2458-13-917. PMID 24088419
- See also: University of Southern Denmark — http://www.sdu.dk